CLINICAL TRIAL: NCT04126486
Title: GUARD-AF: reducinG Stroke by Screening for UndiAgnosed atRial Fibrillation in Elderly inDividuals
Brief Title: A Study to Determine if Identification of Undiagnosed Atrial Fibrillation in People at Least 70 Years of Age Reduces the Risk of Stroke
Acronym: GUARD-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV185-749
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zio®XT Monitor Arm (Other)
  Interventions: Other: Zio®XT Monitor
- Usual Care Arm (No Intervention)

INTERVENTIONS:
Other: Zio®XT Monitor — A Zio® XT monitor will be affixed to the participant's chest
  Arms: Zio®XT Monitor Arm

SUMMARY:
The purpose of this study is to determine if an AF detection intervention in men and women at least 70 years of age with undiagnosed atrial fibrillation (AF) or atrial flutter (AFL) reduces the person-years incidence rate of stroke compared to usual care (no AF detection intervention).

DETAILED DESCRIPTION:
This a prospective, randomized study in primary care practices.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 70 years of age who are new or established participants in the primary care practice
* Willing to provide consent to participate in the study and to use personal health information to ascertain endpoints from the Center for Medicare & Medicaid Services (CMS) Medicare Claims Database and to access data from health records
* Health insurance by Medicare Parts A & B (Medicare Fee-for-service)

Exclusion Criteria:

* Oral anticoagulation (OAC) for any indication at the time of enrollment
* History of Atrial Fibrillation (AF) or Atrial Flutter (AFL) as documented in the participant's current medical problem list
* Any condition the investigator considers a contraindication to OAC, e.g., bleeding that required medical attention or severe renal impairment
* Any condition the investigator considers will prevent compliance with study instructions
* Implanted cardiac devices (pacemakers, implantable cardiac defibrillators, or cardiac resynchronization therapy, and implantable loop recorders)
* History of allergy to adhesive
* Not able to wear the Zio®XT monitor or not able to apply the monitor by herself/himself or with the help of a caregiver

Other protocol-defined inclusion/exclusion criteria could apply

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11931 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of all strokes leading to hospitalization | From 2.5 years to 5 years after study start
Incidence of bleeding leading to hospitalization | From 2.5 years to 5 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (174):
- United States (174):
  - Local Institution - 0302, Birmingham, Alabama
  - Local Institution - 0360, Guntersville, Alabama
  - Local Institution - 0158, Montgomery, Alabama
  - Local Institution - 0109, Kingman, Arizona
  - Local Institution - 0047, Peoria, Arizona
  - Local Institution - 0237, Peoria, Arizona
  - Local Institution - 0171, Phoenix, Arizona
  - Local Institution - 0271, Phoenix, Arizona
  - Local Institution - 0323, Yuma, Arizona
  - Local Institution - 0097, Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - Local Institution - 0173, Fremont, California
  - Local Institution - 0110, Fullerton, California
  - Local Institution - 0301, Oakland, California
  - Local Institution - 0248, Sacramento, California
  - Local Institution - 0061, Toluca Lake, California
  - Local Institution, Aventura, Florida
  - Local Institution - 0143, Boynton Beach, Florida
  - Local Institution - 0232, Clearwater, Florida
  - Local Institution - 0017, Clearwater, Florida
  - Local Institution - 0062, DeLand, Florida
  - University Clinical Research-Deland LLC dba Accel Research Sites, DeLand, Florida
  - Local Institution - 0350, Doral, Florida
  - Local Institution - 0367, Fort Lauderdale, Florida
  - Local Institution - 0161, Fort Lauderdale, Florida
  - Vanguard Clinical Research, LLC, Fort Myers, Florida
  - Finlay Medical Research Corp, Greenacres City, Florida
  - Local Institution - 0348, Hialeah, Florida
  - Local Institution - 0358, Hialeah, Florida
  - Local Institution - 0219, Hialeah, Florida
  - Local Institution - 0366, Jacksonville, Florida
  - Local Institution - 0368, Jacksonville, Florida
  - Local Institution - 0277, Jacksonville, Florida
  - Local Institution - 0375, Lake City, Florida
  - Nova Clinical Research Center Inc, Miami, Florida
  - Local Institution - 0025, Miami, Florida
  - Local Institution - 0296, Miami, Florida
  - Local Institution, Miami, Florida
  - Local Institution - 0300, Miami, Florida
  - Local Institution - 0371, Miami, Florida
  - Local Institution - 0149, Miami Beach, Florida
  - Local Institution - 0374, Miami Lakes, Florida
  - Local Institution - 0372, Miami Shores, Florida
  - Local Institution - 0010, Mt. Dora, Florida
  - Local Institution - 0058, Oviedo, Florida
  - Local Institution - 0132, Palm Harbor, Florida
  - Local Institution - 0034, Palm Springs, Florida
  - Local Institution - 0028, Tampa, Florida
  - Local Institution - 0090, Tampa, Florida
  - Local Institution - 0361, Weston, Florida
  - Local Institution - 0263, Albany, Georgia
  - Local Institution - 0027, Atlanta, Georgia
  - Local Institution, Columbus, Georgia
  - Local Institution - 0033, Eatonton, Georgia
  - Local Institution - 0176, Fayetteville, Georgia
  - Local Institution - 0214, Rincon, Georgia
  - Local Institution - 0098, Savannah, Georgia
  - Local Institution - 0123, Woodstock, Georgia
  - Local Institution - 0311, Chicago, Illinois
  - Local Institution - 0345, Evergreen Park, Illinois
  - Local Institution - 0241, Gillespie, Illinois
  - Local Institution - 0306, Wauconda, Illinois
  - Local Institution - 0365, Indianapolis, Indiana
  - Local Institution - 0254, Michigan City, Indiana
  - Local Institution - 0338, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - Local Institution - 0244, Wichita, Kansas
  - Local Institution - 0369, Lexington, Kentucky
  - Local Institution - 0133, Eunice, Louisiana
  - Local Institution - 0321, New Orleans, Louisiana
  - Local Institution - 0229, Zachary, Louisiana
  - Local Institution - 0351, Annapolis, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Local Institution - 0037, Elkridge, Maryland
  - Local Institution - 0095, Rockville, Maryland
  - Local Institution - 0284, Boston, Massachusetts
  - Local Institution - 0051, Boston, Massachusetts
  - Local Institution - 0333, Haverhill, Massachusetts
  - Local Institution - 0201, New Bedford, Massachusetts
  - Local Institution - 0227, Worcester, Massachusetts
  - Local Institution - 0260, Caro, Michigan
  - Local Institution - 0005, Detroit, Michigan
  - Local Institution - 0166, Sterling Heights, Michigan
  - Local Institution - 0257, Troy, Michigan
  - Local Institution - 0256, Rochester, Minnesota
  - Belzoni Family Practice, Belzoni, Mississippi
  - Local Institution - 0089, Jackson, Mississippi
  - Local Institution - 0224, Petal, Mississippi
  - Local Institution - 0060, Picayune, Mississippi
  - Quinn Healthcare/SKYCRNG, Ridgeland, Mississippi
  - Local Institution - 0116, St Louis, Missouri
  - Local Institution - 0063, Norfolk, Nebraska
  - Local Institution - 0222, Henderson, Nevada
  - Local Institution, Las Vegas, Nevada
  - Local Institution - 0334, Linden, New Jersey
  - Local Institution - 0249, Brooklyn, New York
  - Local Institution - 0362, Cooperstown, New York
  - Local Institution, East Syracuse, New York
  - Local Institution - 0102, Endwell, New York
  - Local Institution - 0379, Niagara Falls, New York
  - Digiovanna Institute For Medical Education, North Massapequa, New York
  - Local Institution, Black Mountain, North Carolina
  - Local Institution - 0328, Burlington, North Carolina
  - Local Institution - 0164, Cary, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Local Institution - 0207, Charlotte, North Carolina
  - Local Institution - 0006, Durham, North Carolina
  - Local Institution, Fayetteville, North Carolina
  - Local Institution - 0268, Franklinton, North Carolina
  - Local Institution - 0258, Greensboro, North Carolina
  - Local Institution - 0159, Hickory, North Carolina
  - Local Institution - 0331, Matthews, North Carolina
  - Local Institution - 0230, Raleigh, North Carolina
  - Local Institution - 0175, Rocky Mount, North Carolina
  - Local Institution - 0253, Salisbury, North Carolina
  - Local Institution - 0153, Statesville, North Carolina
  - Local Institution - 0182, Statesville, North Carolina
  - Local Institution - 0235, Wilmington, North Carolina
  - Local Institution - 0167, Winston-Salem, North Carolina
  - Sterling Research Group, Cincinnati, Ohio
  - Local Institution - 0085, Cincinnati, Ohio
  - Local Institution - 0283, Cleveland, Ohio
  - Local Institution - 0036, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Local Institution - 0212, Dayton, Ohio
  - Local Institution - 0129, Philadelphia, Pennsylvania
  - Local Institution - 0272, Pittsburgh, Pennsylvania
  - Local Institution - 0236, Pittsburgh, Pennsylvania
  - Local Institution - 0349, Pittsburgh, Pennsylvania
  - Local Institution - 0347, Uniontown, Pennsylvania
  - Local Institution - 0370, Uniontown, Pennsylvania
  - Local Institution - 0240, East Providence, Rhode Island
  - Local Institution - 0155, Bristol, Tennessee
  - Local Institution - 0234, Knoxville, Tennessee
  - Local Institution - 0324, Morristown, Tennessee
  - Local Institution - 0309, Nashville, Tennessee
  - Wellness Clinical Research, Allen, Texas
  - Local Institution - 0187, Austin, Texas
  - Local Institution - 0243, Austin, Texas
  - HRMD Research, Dallas, Texas
  - Local Institution - 0242, Denton, Texas
  - Invesclinic.U.S,LLC, Edinburg, Texas
  - Local Institution - 0141, Friendswood, Texas
  - Local Institution - 0354, Georgetown, Texas
  - Local Institution - 0011, Houston, Texas
  - Local Institution - 0343, Houston, Texas
  - Local Institution - 0016, Hurst, Texas
  - Local Institution - 0151, Laredo, Texas
  - Local Institution - 0170, Mesquite, Texas
  - Local Institution - 0101, Pearland, Texas
  - Local Institution - 0223, Pflugerville, Texas
  - Local Institution - 0303, Pharr, Texas
  - Local Institution - 0204, Plano, Texas
  - Local Institution - 0067, Plano, Texas
  - SA Premiere Internal Medicine, San Antonio, Texas
  - Local Institution - 0092, San Antonio, Texas
  - Local Institution - 0278, San Marcos, Texas
  - Local Institution - 0055, Sugar Land, Texas
  - Local Institution - 0137, Sugar Land, Texas
  - Local Institution - 0251, The Woodlands, Texas
  - Local Institution - 0147, The Woodlands, Texas
  - Local Institution - 0322, Tyler, Texas
  - Local Institution - 0150, Bountiful, Utah
  - Local Institution - 0339, Appomattox, Virginia
  - Local Institution - 0191, Burke, Virginia
  - Local Institution - 0340, Forest, Virginia
  - Local Institution - 0267, Suffolk, Virginia
  - Local Institution - 0096, Winchester, Virginia
  - Local Institution - 0364, Winchester, Virginia
  - Local Institution - 0086, Everett, Washington
  - Local Institution - 0299, Tacoma, Washington
  - Local Institution - 0337, Eau Claire, Wisconsin
  - Local Institution - 0335, La Crosse, Wisconsin
  - Local Institution - 0288, Madison, Wisconsin

REFERENCES:
- [Derived] Singer DE, Atlas SJ, Go AS, Lubitz SA, McManus DD, Dolor RJ, Chatterjee R, Rothberg MB, Rushlow DR, Crosson LA, Aronson RS, Mills D, Patlakh M, Gallup D, O'Brien EC, Lopes RD. Atrial Fibrillation Burden on a 14-Day ECG Monitor: Findings From the GUARD-AF Trial Screening Arm. JACC Clin Electrophysiol. 2025 Jan;11(1):110-119. doi: 10.1016/j.jacep.2024.08.010. Epub 2024 Sep 1. PMID 39297839
- [Derived] Lopes RD, Atlas SJ, Go AS, Lubitz SA, McManus DD, Dolor RJ, Chatterjee R, Rothberg MB, Rushlow DR, Crosson LA, Aronson RS, Patlakh M, Gallup D, Mills DJ, O'Brien EC, Singer DE. Effect of Screening for Undiagnosed Atrial Fibrillation on Stroke Prevention. J Am Coll Cardiol. 2024 Nov 19;84(21):2073-2084. doi: 10.1016/j.jacc.2024.08.019. Epub 2024 Sep 1. PMID 39230544
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html